CLINICAL TRIAL: NCT03738527
Title: Pilot RCT: Use of Tranexamic Acid (TXA) in Post Mastectomy Patients for Seroma and Hematoma Prevention
Brief Title: SEroma Reduction pOst MAstectomy "SEROMA Study"
Acronym: SEROMA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5271
Record Dates: First submitted 2018-10-11; First posted 2018-11-13 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Seroma Complicating A Procedure; Hematoma Postoperative; Breast Cancer
Keywords: tranexamic acid; mastectomy; topical; breast cancer; seroma; hematoma
MeSH Terms: conditions — Breast Neoplasms; Seroma; Hematoma | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Pilot Randomized Controlled Trial (RCT) with 2 arms: the interventional arm (receiving topical TXA) and the control arm (receiving placebo).
  Intervention: Topical application of 20 mL of TXA (100 mg/mL injection solution) to the mastectomy cavity
  Placebo: Topical application of 20 mL of 0.9% NaCl (normal saline) to the mastectomy cavity
Who Masked: Participant, Care Provider
Masking Description: Patients will be randomized on the REDCap system. Their assignment will be made available to pharmacy, which will be prepare syringes with either TXA or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TXA arm (Experimental)
  Interventions: Drug: Tranexamic Acid 100mg/mL, 20mL topical
- Placebo arm (Placebo Comparator)
  Interventions: Drug: Normal Saline Flush, 0.9%, 20mL topical

INTERVENTIONS:
Drug: Tranexamic Acid 100mg/mL, 20mL topical — Drug: Tranexamic Acid
  20 mL TXA (100 mg/mL injection solution, total 2g TXA) applied topically to the mastectomy cavity for 5 minutes before wound closure
  Arms: TXA arm
Drug: Normal Saline Flush, 0.9%, 20mL topical — Drug: Normal Saline
  20 mL 0.9% NaCl (normal saline) applied topically to the mastectomy cavity for 5 minutes before wound closure
  Arms: Placebo arm

SUMMARY:
This is a pilot study to evaluate the feasibility of conducting a larger trial to determine if the use of intraoperative topical tranexamic acid (TXA) decreases the rate of post-operative hematomas and seromas in breast cancer patients after their mastectomy. In other words, the investigators want to determine if applying TXA inside the surgical wound before it is closed helps reduce blood or serous fluid accumulation at the operative site. Dependent on the results of this study, a further larger trial may or may not take place.

Post-operative seromas and hematomas are common complications of mastectomy surgery not only leading to infection, discomfort, wound dehiscence or emergency room visits; they also delay in some instances post-operative adjuvant radiotherapy. Establishing whether or not topical TXA is an effective strategy to decrease those complications can potentially impact positively the breast cancer treatment.

To achieve this aim, this randomized pilot study will first determine whether a larger multicenter study if feasible. This study will replicate a formal randomized trial at a smaller scale in a single center in order to assess the recruitment and randomization process, as well as provide preliminary results for our research question.

DETAILED DESCRIPTION:
The objective of this study is to investigate the novel use of topical application of Tranexamic Acid (TXA) to the surgical wound as a means to decrease seroma and/or hematoma formation compared to placebo in post-mastectomy patients. This project is designed as a single-center pilot RCT to evaluate the feasibility of conducting a formal RCT (multicenter trial including more patients) to evaluate the effectiveness of topical TXA.

Patients will be randomly assigned to one of two treatment groups for intraoperative treatment of their mastectomy wound before it is closed.

The first group will consist of those who will be treated with the intravenous form of TXA that will be applied to the surface of the mastectomy wound area rather than being injected into a vein. The second group consists of those individuals who will be treated with a topical normal saline solution (a placebo, or inactive substance that looks identical to the study drug but contains no therapeutic ingredients).

Both groups will receive the same number of drains and the same post-operative follow-up schedule consisting of visits 2 to 4 weeks and 3 months after the surgery, as well as a last 12 months follow-up. Standard of care will be practiced with respect to all procedures and visits.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosis
* Age 18-80
* Fluent in English
* Female undergoing mastectomy with or without axillary intervention

Exclusion Criteria:

* Immediate reconstruction
* Pre-surgical radiation
* Known allergy to TXA
* Known thromboembolic disease
* High-risk of thromboembolism and/or receiving anticoagulants
* History of myocardial infarction (MI), transient ischemic attack or stroke within the last year
* History of subarachnoid hemorrhage
* Premenopausal women with irregular menstrual bleeding of unknown cause
* Acquired disturbances of colour vision
* Hematuria with renal cause
* History of seizure disorder
* Pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | About 6 months
  Number of patients recruited over the total number of eligible patients screened
Randomization rate | About 9 months
  Number of patients randomized over total number recruited
Follow-up visit rate | 3 months
  Number of patients with successful follow-up visits at 3 weeks and 3 months
Ability to adhere to protocol | About 12 months
  Number of patients randomized to TXA who received TXA vs number of patients randomized to placebo who received the placebo

SECONDARY OUTCOMES:
Seroma rate | 3 months
  Rate of seroma formation within 3 months following mastectomy in each arm of the study.
Seroma volume | 3 months
  Amount of drainage (volume) in patients who did have a seroma, for patients in both arms of the study
Seroma aspiration | 3 months
  Aspirated volume in patients who did have a seroma, for patients in both arms of the study
Delay in adjuvant treatment | 3 months
  Time (number of weeks) of delay in adjuvant treatment due to seroma/hematoma complication, for patients in both arms of the study

OTHER OUTCOMES:
Other complications rate: Hematoma rate | 3 months
  Rate of hematoma within 3 months following mastectomy in each arm of the study
Other complications rate: Infection rate | 3 months
  Rate of infection within 3 months following mastectomy in each arm of the study
Other complications rate: Wound dehiscence rate | 3 months
  Rate of wound dehiscence within 3 months following mastectomy in each arm of the study
Daily output volume | 3 months
  Daily drain output (volume), in patients in both arms of the study
Drain discontinuation | 3 months
  Time to drain discontinuation (number of days) in patients in both arms of the study
Drain complications | 3 months
  Presence of drain complications (leakage, dislodgement, blockage), in patients in both arms of the study
Safety outcomes: rate of thromboembolic events | 3 weeks
  Rate of Thromboembolic events within 3 weeks following mastectomy, in patients in both arms of the study
Safety outcomes: rate of myocardial events | 3 weeks
  Rate of myocardial events within 3 weeks following mastectomy, in patients in both arms of the study
  • Rate of other adverse events within 3 weeks following mastectomy
Safety outcomes: rate of other adverse events | 3 weeks
  Rate of other adverse events within 3 weeks following mastectomy, in patients in both arms of the study

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Hodgson, MD, MSc, FRCSC, Principal Investigator — Hamilton Health Sciences, McMaster University
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Hospital - Hamilton Health Sciences, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porter KA, O'Connor S, Rimm E, Lopez M. Electrocautery as a factor in seroma formation following mastectomy. Am J Surg. 1998 Jul;176(1):8-11. doi: 10.1016/s0002-9610(98)00093-2. PMID 9683123
- [Background] Pogson CJ, Adwani A, Ebbs SR. Seroma following breast cancer surgery. Eur J Surg Oncol. 2003 Nov;29(9):711-7. doi: 10.1016/s0748-7983(03)00096-9. PMID 14602488
- [Background] van Bemmel AJ, van de Velde CJ, Schmitz RF, Liefers GJ. Prevention of seroma formation after axillary dissection in breast cancer: a systematic review. Eur J Surg Oncol. 2011 Oct;37(10):829-35. doi: 10.1016/j.ejso.2011.04.012. Epub 2011 Aug 17. PMID 21849243
- [Background] Coveney EC, O'Dwyer PJ, Geraghty JG, O'Higgins NJ. Effect of closing dead space on seroma formation after mastectomy--a prospective randomized clinical trial. Eur J Surg Oncol. 1993 Apr;19(2):143-6. PMID 8491318
- [Background] Baker E, Piper J. Drainless mastectomy: Is it safe and effective? Surgeon. 2017 Oct;15(5):267-271. doi: 10.1016/j.surge.2015.12.007. Epub 2016 Feb 19. PMID 26907221
- [Background] He XD, Guo ZH, Tian JH, Yang KH, Xie XD. Whether drainage should be used after surgery for breast cancer? A systematic review of randomized controlled trials. Med Oncol. 2011 Dec;28 Suppl 1:S22-30. doi: 10.1007/s12032-010-9673-2. Epub 2010 Sep 9. PMID 20827578
- [Background] Ker K, Roberts I, Shakur H, Coats TJ. Antifibrinolytic drugs for acute traumatic injury. Cochrane Database Syst Rev. 2015 May 9;2015(5):CD004896. doi: 10.1002/14651858.CD004896.pub4. PMID 25956410
- [Background] Gupta K, Rastogi B, Krishan A, Gupta A, Singh VP, Agarwal S. The prophylactic role of tranexamic acid to reduce blood loss during radical surgery: A prospective study. Anesth Essays Res. 2012 Jan-Jun;6(1):70-3. doi: 10.4103/0259-1162.103378. PMID 25885506
- [Background] Perel P, Ker K, Morales Uribe CH, Roberts I. Tranexamic acid for reducing mortality in emergency and urgent surgery. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD010245. doi: 10.1002/14651858.CD010245.pub2. PMID 23440847
- [Background] Oertli D, Laffer U, Haberthuer F, Kreuter U, Harder F. Perioperative and postoperative tranexamic acid reduces the local wound complication rate after surgery for breast cancer. Br J Surg. 1994 Jun;81(6):856-9. doi: 10.1002/bjs.1800810621. PMID 8044602
- [Background] Ker K, Beecher D, Roberts I. Topical application of tranexamic acid for the reduction of bleeding. Cochrane Database Syst Rev. 2013 Jul 23;2013(7):CD010562. doi: 10.1002/14651858.CD010562.pub2. PMID 23881695
- [Background] Xu X, Xiong S, Wang Z, Li X, Liu W. Topical administration of tranexamic acid in total hip arthroplasty: A meta-analysis of Randomized Controlled Trials. Drug Discov Ther. 2015 Jun;9(3):173-7. doi: 10.5582/ddt.2015.01018. PMID 26193938
- [Background] Ausen K, Fossmark R, Spigset O, Pleym H. Randomized clinical trial of topical tranexamic acid after reduction mammoplasty. Br J Surg. 2015 Oct;102(11):1348-53. doi: 10.1002/bjs.9878. PMID 26349843
- [Background] Bennett C, Klingenberg SL, Langholz E, Gluud LL. Tranexamic acid for upper gastrointestinal bleeding. Cochrane Database Syst Rev. 2014 Nov 21;2014(11):CD006640. doi: 10.1002/14651858.CD006640.pub3. PMID 25414987